CLINICAL TRIAL: NCT04125758
Title: Is Knowing the Body Knowing the Mind? Stress-physiology Coherence, Interoception, and Mindfulness
Brief Title: Stress-physiology Coherence, Interoception, and Well-being Following Mindfulness Training or Tracking Time Spent on Mobile Device
Acronym: SCIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-0153; A487400 (Other: UW Madison); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW Madison); Protocol Version 6/10/2022 (Other: UW Madison)
Record Dates: First submitted 2019-09-05; First posted 2019-10-14 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Not Seeking to Treat Any Conditions
MeSH Terms: interventions — Mindfulness; Meditation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned after a baseline testing to either a mindfulness intervention or control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers involved in participant testing will not know the participant's group. Researchers conducting data analysis will not know data codes assigned to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (Experimental): Participants will listen to one to two 3-30 minute audio recordings each day for 4 weeks between study visits (28 days total) through the Healthy Minds @Work smartphone app and record when they listen to each recording on a paper log. The app will also collect data on which recordings, when, and for how long participants listen.
  Interventions: Behavioral: Mindfulness training
- Tracking time spent on mobile device (Active Comparator): Participants will record how much time they estimate they have spent on their phone in the past 24 hours, each day for 4 weeks (28 days total) between study visits.
  Interventions: Behavioral: Tracking time spent on mobile device

INTERVENTIONS:
Behavioral: Mindfulness training — Brief audio recordings discussing mindfulness or guided mindfulness practices.
  Other Names: Mindfulness, contemplative, meditation
  Arms: Mindfulness training
Behavioral: Tracking time spent on mobile device — Participants will record each day how much time they estimate they spent on their smart phone in the past 24 hours.
  Arms: Tracking time spent on mobile device

SUMMARY:
Chronic stress has been shown to impact long-term emotional and physical health. When nearly three-quarters of Americans report stress at levels that exceed what they consider healthy, there is a desperate need to understand factors that contribute to effective stress regulation. This work seeks to develop a measure tied to awareness and acceptance of stress that has shown promise as a predictor of multiple markers of mental and physical well-being, understand how it relates to awareness of the body, and explore whether it can be trained to alleviate suffering and promote well-being. This study aims to 1) Conceptually replicate and extend previous findings linking greater stress-physiology coherence to higher well-being. 2) Assess whether awareness of physiology is associated with stress-physiology coherence. 3) Explore whether stress-physiology coherence can be trained through a brief mindfulness training intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65;
2. Comfortable reading, writing, and conversing in English
3. U.S. Citizen or permanent resident (for payment purposes)
4. Have a smartphone compatible with our study app

Exclusion Criteria:

1. Significant past experience with meditation, yoga, tai chi, or qi gong;
2. Current or past psychotic disorder, Bipolar Disorder, PTSD, or social phobia;
3. Current, severe major depressive episode;
4. Current, severe generalized anxiety;
5. Active prescription stimulant use (current or in the past month);
6. Active prescription beta-blocker, beta-agonist, anti-high blood pressure, or anti-anxiety medication use (current or in the past month);
7. Currently pregnant (due to physiological changes);
8. History of neurological disorder;
9. Currently diagnosed with high blood pressure, or heart murmur;
10. Have a pacemaker
11. Have participated in the Trier Social Stress Test previously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in subjective stress-heart rate coherence | Baseline and post-test, separated by 4 weeks
  Within-participant association between repeated measures of subjective stress (1-100 Visual Analog Scale rating) and heart rate over the course of a stress-induction paradigm. Stronger positive associations indicate higher stress-heart rate coherence.

OTHER OUTCOMES:
Mean Change in Accuracy on Method of Constant Stimuli (MCS) Interoceptive Accuracy Task | Baseline and post-test, separated by 4 weeks
  Participants will complete a modified version of the MCS heart beat detection task used by Brener, Ring, and Liu. Participants will be asked to report whether a series of five tones are simultaneous with five of their heart beats. Each trial involves five heart beats. Each heart beat is followed by a tone, and the lag between heart beat and tone is varied across trials with five delay conditions: 0 ms, 100 ms, 200 ms, 300 ms, 400 ms, or 500 ms. Thus, each trial involves five beat-tone pairs, separated according to a single delay condition. Delays will be pseudorandomly presented across trials. Varying delays allow for individual differences in when participants perceive their heart beat. A continuous measure of judgement precision is defined as the participant's interquartile range (IQR) of the distribution of percent of simultaneous responses for each delay condition. IQR ranges from 0 to 450. Lower IQRs indicate more consistent responses and thus higher accuracy.
Mean Change in Interoceptive Sensibility measured as the total score on the Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2) | Baseline and post-test, separated by 4 weeks
  Interoceptive Sensibility measured as the total score on the Multidimensional Assessment of Interoceptive Awareness Version 2. Scores range from 0 to 185. Higher scores indicate greater interoceptive sensibility.
Mean Change in Meta-Awareness Measured on a Method of Constant Stimuli Light-Tone Task | Baseline and post-test, separated by 4 weeks
  Participants will complete a Method of Constant Stimuli (MCS) light-tone task. Participants will be asked to report whether a series of five tones are simultaneous with five light flashes. Each trial involves five light-tone pairs. Each light flash is followed by a tone, and the lag between light flash and tone is varied across trials with five delay conditions: 0 ms, 100 ms, 200 ms, 300 ms, 400 ms, or 500 ms. Thus, each trial involves five light-tone pairs, separated according to a single delay condition. Delays will be pseudorandomly presented across trials. After each trial in the task, participants will be asked how confident they are in their response on a simple likert scale ranging from 1 = not at all confident to 4 = completely confident. Meta-awareness is defined as the correlation between accurate responses (simultaneous judgements at the 0 ms delay) and confidence ratings. Scores thus range from -1 to 1. Higher scores indicate more meta-awareness.
Mean Change in Total (Sum) Score on the Cognitive Fusion Questionnaire (CFQ) | Baseline and post-test, separated by 4 weeks
  Cognitive Fusion Questionnaire (CFQ) total (sum) score. Scores range from 7-49. Greater numbers reflect greater cognitive fusion.
Mean Change in Internal Locus of Control Subscale Total (Sum) Score of the Locus of Control (LOC) | Baseline and post-test, separated by 4 weeks
  Internal locus of control subscale total (sum) score of the Locus of Control (LOC). Scores range from 0-48 on this subscale. Higher scores indicate greater internal locus of control.
Mean Change in Total (Sum) Score on Psychological Well Being Scale (42-item version) | Baseline and post-test, separated by 4 weeks
  Total score (sum) on Psychological Well Being Scale (42-item version). Scores range from 42 to 294. Higher scores indicate higher psychological well-being.
Mean Change in Total (Sum) Score on the Brief Experiential Avoidance Questionnaire (BEAQ) | Baseline and post-test, separated by 4 weeks
  Brief Experiential Avoidance Questionnaire (BEAQ) total (sum) score. Scores ranger from 15 to 90. Higher scores indicate greater experiential avoidance.
Mean Change in Acceptance Subscale Total (Sum) Score of the COPE Questionnaire | Baseline and post-test, separated by 4 weeks
  Acceptance subscale total (sum) score of the COPE questionnaire. Scores range from 4 to 16. Higher scores indicate more use of acceptance coping.
Mean Change in Denial Subscale Total (Sum) Score of the COPE Questionnaire | Baseline and post-test, separated by 4 weeks
  Denial subscale total (sum) score of the COPE questionnaire. Scores range from 4 to 16. Higher scores indicate more use of denial coping.
Mean Change in Total (Sum) Score on Center for Epidemiological Studies Depression Inventory - Revised 20-item (CESD-R-20) | Baseline and post-test, separated by 4 weeks
  Total score (sum) on Center for Epidemiological Studies Depression Inventory - Revised 20-item. Scores range from 0 to 60, with higher scores indicating more depressive symptoms.
Mean Change in Total (Sum) Score on Spielberger Trait Anxiety Inventory Y2 | Baseline and post-test, separated by 4 weeks
  Total (Sum) Score on Spielberger Trait Anxiety Inventory Y2. Scores range from 20-80. Higher scores indicate greater trait anxiety.
Mean Change in Global Score on Pittsburgh Sleep Quality Index (PSQI) | Baseline and post-test, separated by 4 weeks
  Global score on Pittsburgh Sleep Quality Index (PSQI). Global scores range from 0 to 21. Higher scores indicate worse sleep quality.
Mean Change in Total (Sum) Score on Perceived Stress Scale-10 (PSS-10) | Baseline and post-test, separated by 4 weeks
  Total (sum) score on Perceived Stress Scale-10 (PSS-10). Scores range from 0 to 40. Higher scores indicating higher perceived stress.
Mean Change in Nonjudging of Inner Experience Subscale Total (Sum) Score on the Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and post-test, separated by 4 weeks
  Nonjudging of Inner Experience Subscale Total (Sum) Score on the Five Facet Mindfulness Questionnaire (FFMQ). Scores on this subscale range from 8-40. Higher scores indicate greater nonjudging of inner experience.
Mean Change in Observing Subscale Total (Sum) Score on the Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and post-test, separated by 4 weeks
  Observing Subscale Total (Sum) Score on the Five Facet Mindfulness Questionnaire (FFMQ). Scores on this subscale range from 8-40. Higher scores indicate greater observing of experience.
Mean Change in Self-Awareness Subscale Total (Sum) Score on the Emotional Styles Questionnaire (ESQ) | Baseline and post-test, separated by 4 weeks
  Self-Awareness Subscale Total (Sum) Score on the Emotional Styles Questionnaire (ESQ). Scores on this subscale range from 4-28. Higher scores indicate greater self-awareness.
Mean Change in Difficulty Identifying Feelings Subscale Total (Sum) Score on the Toronto Alexithymia Scale (TAS-20) | Baseline and post-test, separated by 4 weeks
  Difficulty Identifying Feelings Subscale Total (Sum) Score on the Toronto Alexithymia Scale (TAS-20; Bagby, Parker, & Taylor, 1994). Scores range from 20-60. Greater scores indicate stronger alexithymia.
Mean Change in Incremental Mindset Total (Average) Score on the Dweck Mindset Instrument (DWI) | Baseline and post-test, separated by 4 weeks
  Scores range from 1 to 6. Lower scores indicate more fixed/entity views of intelligence and talent. Higher scores indicate more incremental/malleable views of intelligence and talent.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Sommerfeldt, M.S., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data only may be banked for future use to address research questions not included in this registration.
  We may share coded data with other researchers within and outside of UW-Madison, and data may also be used in additional future approved research studies. These studies may include analysis of the information from this study alone or in combination with data collected in other studies.
  All data except Protected Health Information may be shared. Data may be shared as Supplemental Information uploaded to a journal website and/or shared on a UW data sharing website. Data sharing would not require any further participation from participants. Participants may withdraw their data from future research by submitting a request in writing to our study team.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after Sasha Sommerfeldt's dissertation defense. The study protocol, analysis plan, informed consent form, and analytic code will be shared publicly through the open science framework upon acceptance of a manuscript detailing findings for the main aims of the study. Data will be shared upon request from qualified researchers.

REFERENCES:
- [Background] Birkett MA. The Trier Social Stress Test protocol for inducing psychological stress. J Vis Exp. 2011 Oct 19;(56):3238. doi: 10.3791/3238. PMID 22042290
- [Background] Ekman, P. (1992). An argument for basic emotions. Cognition & emotion, 6(3-4), 169-200.
- [Background] Mauss IB, Levenson RW, McCarter L, Wilhelm FH, Gross JJ. The tie that binds? Coherence among emotion experience, behavior, and physiology. Emotion. 2005 Jun;5(2):175-90. doi: 10.1037/1528-3542.5.2.175. PMID 15982083
- [Background] Campbell J, Ehlert U. Acute psychosocial stress: does the emotional stress response correspond with physiological responses? Psychoneuroendocrinology. 2012 Aug;37(8):1111-34. doi: 10.1016/j.psyneuen.2011.12.010. Epub 2012 Jan 18. PMID 22260938
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Darwin, C. (2009). The expression of the emotions in man and animals (P. Ekman, Ed.). Oxford, England: Oxford University Press. (Original work published 1872)
- [Background] Garfinkel SN, Manassei MF, Hamilton-Fletcher G, In den Bosch Y, Critchley HD, Engels M. Interoceptive dimensions across cardiac and respiratory axes. Philos Trans R Soc Lond B Biol Sci. 2016 Nov 19;371(1708):20160014. doi: 10.1098/rstb.2016.0014. Epub 2016 Oct 10. PMID 28080971
- [Background] Hirshberg MJ, Goldberg SB, Schaefer SM, Flook L, Findley D, Davidson RJ. Divergent effects of brief contemplative practices in response to an acute stressor: A randomized controlled trial of brief breath awareness, loving-kindness, gratitude or an attention control practice. PLoS One. 2018 Dec 12;13(12):e0207765. doi: 10.1371/journal.pone.0207765. eCollection 2018. PMID 30540772
- [Background] Lang, P. J. (1988). What are the data of emotion? In V. Hamilton, G. H. Bower, & N. Frijda (Eds.), Cognitive perspectives on emotion and motivation (pp. 173-191). Amsterdam, The Netherlands: Martinus Nijhoff Publishers.
- [Background] Lazarus, R. S. (1991). Emotion and adaptation. Oxford, England: Oxford University Press.
- [Background] Levenson, R. W. (1994). Human emotion: A functional view. In P. Ekman & R. J. Davidson (Eds.), The nature of emotion: Fundamental questions (pp. 123-126). New York, NY: Oxford University Press.
- [Background] Plutchik, R. (1980). Emotion: A psychoevolutionary synthesis. New York, NY: HarperCollins College Division.
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied Psychology Measurement, 1, 385-401.
- [Background] Ryff, C. D. (1989). Happiness is everything, or is it? Explorations on the meaning of psychological well-being. Journal of Personality and Social Psychology, 57, 1069-1081.
- [Background] Sommerfeldt SL, Schaefer SM, Brauer M, Ryff CD, Davidson RJ. Individual Differences in the Association Between Subjective Stress and Heart Rate Are Related to Psychological and Physical Well-Being. Psychol Sci. 2019 Jul;30(7):1016-1029. doi: 10.1177/0956797619849555. Epub 2019 Jun 12. PMID 31188735
- [Background] Spielberger, C. D. (1983). Manual for the State-Trait Anxiety Inventory (Form Y) ("Self-Evaluation Questionnaire"). Palo Alto, CA: Consulting Psychologists Press.
- [Background] Sze JA, Gyurak A, Yuan JW, Levenson RW. Coherence between emotional experience and physiology: does body awareness training have an impact? Emotion. 2010 Dec;10(6):803-14. doi: 10.1037/a0020146. PMID 21058842
- [Background] Brener J, Ring C, Liu X. Effects of data limitations on heartbeat detection in the method of constant stimuli. Psychophysiology. 1994 May;31(3):309-12. doi: 10.1111/j.1469-8986.1994.tb02219.x. PMID 8008794
- [Background] Brener J, Liu X, Ring C. A method of constant stimuli for examining heartbeat detection: comparison with the Brener-Kluvitse and Whitehead methods. Psychophysiology. 1993 Nov;30(6):657-65. doi: 10.1111/j.1469-8986.1993.tb02091.x. PMID 8248457
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Levenson H. Multidimensional locus of control in psychiatric patients. J Consult Clin Psychol. 1973 Dec;41(3):397-404. doi: 10.1037/h0035357. No abstract available. PMID 4803272
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Kesebir P, Gasiorowska A, Goldman R, Hirshberg MJ, Davidson RJ. Emotional Style Questionnaire: A multidimensional measure of healthy emotionality. Psychol Assess. 2019 Oct;31(10):1234-1246. doi: 10.1037/pas0000745. Epub 2019 Jul 1. PMID 31259572
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474